CLINICAL TRIAL: NCT02674594
Title: An Early Evaluation of 30-Day Readmissions Among Nonvalvular Atrial Fibrillation (NVAF) Patients Treated With Dabigatran, Rivaroxaban, Apixaban, or Warfarin in the US
Brief Title: Evaluation of Hospital Readmissions Among Hospitalized Non-valvular Atrial Fibrillation (NVAF) Patients in the US
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-405
Record Dates: First submitted 2016-01-15; First posted 2016-02-04 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Nonvalvular Atrial Fibrillation
Keywords: Anticoagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patient treated with Dabigatran
- Patient treated with Rivaroxaban
- Patient treated with Apixaban
- Patient treated with Warfarin

SUMMARY:
The overall objective of this proposal is to execute a real-world database analysis to evaluate hospital readmissions among hospitalized nonvalvular atrial fibrillation (NVAF) patients in the U.S

Primary objective: To determine the proportions of NVAF patients with bleeding-related hospital readmissions that occur within 30 days of the hospitalization of NVAF patients treated with the new oral anticoagulants (NOACs), dabigatran, rivaroxaban, apixaban or warfarin in the inpatient setting

Secondary objectives:

* To determine the cost associated with bleeding-related hospital readmissions that occur within 30 days of the hospitalization of NVAF patients treated with dabigatran, rivaroxaban, apixaban or warfarin in the inpatient setting
* To determine the proportions of NVAF patients with all cause hospital readmissions and the associated costs that occur within 30 days of the hospitalization of NVAF patients treated with dabigatran, rivaroxaban, apixaban or warfarin in the inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary or secondary diagnosis of AF identified by International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) codes from the Premier Hospital database between January 1, 2012 and December 31, 2013
* Age 18 years or older as of initial hospitalization with AF diagnosis

Exclusion Criteria:

* Have any primary or secondary diagnosis code or procedure code for valvular disease during the study period. This exclusion criterion is consistent with that used in other previous BMS HEOR studies and is used to ensure that the study populations are NVAF patients
* Received multiple types of NOACs during the index hospitalization. Preliminary analysis showed that very few patients receive multiple types of new oral anticoagulants (NOACs) during the same hospitalization. This exclusion criterion will allow to cleanly group patients into the different NOAC usage groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Premier Hospital database is the source of all data
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Proportions of NVAF patients with bleeding related hospital readmissions that occur within 30 days of the hospitalization of NVAF patients treated with the NOACs, dabigatran, rivaroxaban, apixaban, or warfarin in the inpatient setting | 30 days post treatment

SECONDARY OUTCOMES:
The cost associated with bleeding-related hospital readmissions that occur within 30 days of the hospitalization of NVAF patients treated with dabigatran, rivaroxaban, apixaban, or warfarin in the inpatient setting | 30 days post treatment
Proportions of NVAF patients with all cause hospital readmissions that occur within 30 days of the hospitalization of NVAF patients treated with dabigatran, rivaroxaban, apixaban or warfarin in the inpatient setting | 30 days post treatment
Associated costs that occur within 30 days of the hospitalization of NVAF patients treated with dabigatran, rivaroxaban, apixaban or warfarin in the inpatient setting | 30 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx